CLINICAL TRIAL: NCT00067873
Title: Exercise Training in Obesity-prone Black and White Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Gary Hunter, PhD, Principle Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BLKWHT (DK49779) (completed); R01DK049779 (NIH)
Record Dates: First submitted 2003-08-29; First posted 2003-09-01 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet; Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diet only (Active Comparator)
  Interventions: Behavioral: Diet
- Diet plus aerobic exercise (Experimental)
  Interventions: Behavioral: Diet; Behavioral: Aerobic exercise
- Diet plus resistance exercise (Experimental)
  Interventions: Behavioral: Diet; Behavioral: Resistance exercise

INTERVENTIONS:
Behavioral: Diet
Behavioral: Aerobic exercise
  Arms: Diet plus aerobic exercise
Behavioral: Resistance exercise
  Arms: Diet plus resistance exercise

SUMMARY:
Overweight premenopausal Black and White women are randomized to either diet-only, diet+aerobic or diet+resistance exercise training. Diet/behavior intervention, with or without the aerobic or resistance exercise training, will be provided throughout the 18 months of study. Major outcomes will include measures of perceived and physiologic difficulty of exercise (cardiac, ventilatory, electromyographic responses to standardized exercise tasks); aerobic fitness; strength fitness; and spontaneous free-living energy expenditure (all derived from doubly labeled water). The results will provide insight into the effectiveness of, and the mechanisms by which, different types of exercise training can improve physical fitness, spontaneous engagement in physical activities of daily living and, in turn, weight-loss maintenance.

DETAILED DESCRIPTION:
Overweight premenopausal Black and White women are randomized to either diet-only, diet+aerobic or diet+resistance exercise training. Diet/behavior intervention, with or without the aerobic or resistance exercise training, will be provided throughout the 18 months of study. Major outcomes will include measures of perceived and physiologic difficulty of exercise (cardiac, ventilatory, electromyographic responses to standardized exercise tasks); aerobic fitness; strength fitness; and spontaneous free-living energy expenditure (all derived from doubly labeled water). The results will provide insight into the effectiveness of, and the mechanisms by which, different types of exercise training can improve physical fitness, spontaneous engagement in physical activities of daily living and, in turn, weight-loss maintenance.

Time of initial weight loss was defined as the time needed to reach the goal of 25 kg/m2 BMI. The women will then be evaluated one year after this time and the amount of weight gain will be determined.

ELIGIBILITY:
* Normoglycemic
* BMI between 27-30
* Non smoker
* Premenopausal
* Physically untrained
* Family history of obesity

Ages: 21 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 231 (Actual)
Dates: Start 2000-12 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | 6 months
Change in weight after initial weight loss | 12 months after initial weight loss (maximum 18 months after randomization)
  Time of initial weight loss determined by days to reach BMI <= 25 (maximum 6 months)

SECONDARY OUTCOMES:
Insulin sensitivity | 6 months post baseline
Insulin sensitivity | 18 months post baseline
Change in visceral fat | 6 months post baseline
Change in visceral fat | 18 months post baseline
Change in cholesterol | 6 months post baseline
Change in cholesterol | 18 months post baseline
Change in triglycerides | 6 months post baseline
Change in triglycerides | 18 months post baseline
Change in resting energy expenditure | 6 months post baseline
Change in resting energy expenditure | 18 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gary R Hunter, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Hunter GR, Fisher G, Neumeier WH, Carter SJ, Plaisance EP. Exercise Training and Energy Expenditure following Weight Loss. Med Sci Sports Exerc. 2015 Sep;47(9):1950-7. doi: 10.1249/MSS.0000000000000622. PMID 25606816
- [Result] Hunter GR, Brock DW, Byrne NM, Chandler-Laney PC, Del Corral P, Gower BA. Exercise training prevents regain of visceral fat for 1 year following weight loss. Obesity (Silver Spring). 2010 Apr;18(4):690-5. doi: 10.1038/oby.2009.316. Epub 2009 Oct 8. PMID 19816413
- [Derived] Bartholomew CL, Martins C, Gower B. The Role of Insulin Sensitivity in Lean Mass Changes During Weight Loss With or Without Exercise. Obesity (Silver Spring). 2025 Nov;33(11):2103-2111. doi: 10.1002/oby.70010. Epub 2025 Sep 2. PMID 40898644
- [Derived] Martins C, Gower BA, Hunter GR. Changes in Trunk, but Not Limb, Lean Body Mass Contribute to Variability in Metabolic Adaptation Following Weight Loss. Obes Sci Pract. 2025 Mar 19;11(2):e70054. doi: 10.1002/osp4.70054. eCollection 2025 Apr. PMID 40110172
- [Derived] Martins C, Gower BA, Hunter GR. Association between Fat-Free Mass Loss after Diet and Exercise Interventions and Weight Regain in Women with Overweight. Med Sci Sports Exerc. 2022 Dec 1;54(12):2031-2036. doi: 10.1249/MSS.0000000000002992. Epub 2022 Jul 8. PMID 35797356
- [Derived] Martins C, Gower BA, Hill JO, Hunter GR. Metabolic adaptation is not a major barrier to weight-loss maintenance. Am J Clin Nutr. 2020 Sep 1;112(3):558-565. doi: 10.1093/ajcn/nqaa086. PMID 32386226
- [Derived] Brock DW, Tompkins CL, Fisher G, Hunter GR. Influence of resting energy expenditure on blood pressure is independent of body mass and a marker of sympathetic tone. Metabolism. 2012 Feb;61(2):237-41. doi: 10.1016/j.metabol.2011.06.019. Epub 2011 Aug 4. PMID 21820136
- [Derived] Brock DW, Chandler-Laney PC, Alvarez JA, Gower BA, Gaesser GA, Hunter GR. Perception of exercise difficulty predicts weight regain in formerly overweight women. Obesity (Silver Spring). 2010 May;18(5):982-6. doi: 10.1038/oby.2009.318. Epub 2009 Oct 8. PMID 19816412